CLINICAL TRIAL: NCT07005050
Title: Renal Pelvic Denervation Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Verve Medical, Inc (Industry)
Collaborators: RQM+ (Industry); Dabl Ltd (Unknown); Medical Labs Memphis - MLM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CP0005
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Uncontrolled Hypertension

STUDY DESIGN:
Intervention Model Description: The study is multi-center, randomized, double-blind and sham-controlled, with sham treated subjects undergoing a procedure that includes use of cystoscopic placement of a guidewire and sheath into one kidney and then the other, to mirror how subjects are treated with RPD.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study involves a hypertension study investigator and an operating endourologist. In the study, the hypertension investigator and their staff will be blinded to treatment through 12 months follow up. Equally, the patient will be blinded to the treatment. Masking will include isolation of medical records from the procedure and sensory isolation of the patient during procedure. All information will become available to the patient and hypertension team after the 12 months follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RPD arm (Experimental): The Verve RPD™ system is used to perform renal pelvic denervation via the urinary collecting system for the treatment of hypertension. The system does so through the delivery of RF energy to the walls of the renal pelvis - delivered via natural orifice through the urinary tract. During the course of the study, patients will be on active medical therapy for their hypertension.
  Interventions: Device: RPD; Drug: Active hypertension medical therapy
- Sham arm (Sham Comparator): Sham procedure will include all steps employed in the renal pelvis denervation with exception of activation of the RPD™ Device. Sham procedure includes advancing guidewire, cystoscope and sheath to position within the renal pelvis, then deploying the RPD™ Device into the renal pelvis (within each kidney), keeping the device in place for 2 minutes (within each kidney) to simulate activation, and then withdrawing the device and sheath. During the course of the study, sham patients will be on active medical therapy for their hypertension.
  Interventions: Drug: Active hypertension medical therapy

INTERVENTIONS:
Device: RPD — Renal Pelvic Denervation
  Arms: RPD arm
Drug: Active hypertension medical therapy — Prespecified two medication regimen for control of hypertension

SUMMARY:
The RPD Pilot trial will evaluate the safety and effectiveness of Verve Medical's RPDTM renal denervation system for hypertensive patients with uncontrolled blood pressure despite use of two medications at a therapeutic dose.

The novelty of the RPDTM system relates to its placement via natural orifice into the renal pelvis (bilaterally) for delivery of radiofrequency energy to ablate the nerves that pass through the outer wall of the renal pelvis, a technique referred to as renal pelvic denervation (RPD).

DETAILED DESCRIPTION:
Hypertensive patients frequently fail to have blood pressure optimally controlled, even with use of multiple medicines. The risk of chronically uncontrolled hypertension are substantial. Several clinical trials demonstrate the potential utility of renal denervation to improve blood pressure control as an adjunct to medications, yet the results of the technology and associated procedures have proven inconsistent. The RICH Pilot trial will evaluate the safety and effectiveness of Verve Medical's RPDTM renal denervation system for hypertensive patients with uncontrolled blood pressure despite use of two medications at a therapeutic dose.

The novelty of the RPDTM system relates to its placement via natural orifice into the renal pelvis (bilaterally) for delivery of radiofrequency energy to ablate the nerves that pass through the outer wall of the renal pelvis, a technique referred to as renal pelvic denervation (RPD).

Safety and effectiveness assessments will include measurement of ambulatory and automated office blood pressure, renal function, procedural complications and all adverse events. These randomized, double-blind, sham-controlled assessments will be conducted 2-, 6- and 12-months following the index procedure. Following completion of the 12-month assessments, sham treated subjects may receive open-label therapy if they meet the original inclusion/exclusion criteria, with all subjects followed for a total of 2 years.

Up until the Month 6 assessment is complete, anti-hypertensive medical therapy is not to be altered unless required by significant worsening of a hypertensive related disease or due to a hypertensive emergency. Following completion of the Month 6 assessments, blinded investigators will be permitted and encouraged to intensify anti-hypertensive medication(s) if clinically indicated, as described further in the protocol. Between years 1 and 2, investigators will continue to be encouraged to intensify anti-hypertensive therapy for subjects not at goal.

ELIGIBILITY:
Inclusion Criteria:

1. Currently taking 2 anti-hypertensive medications (NOTE: no changes to medications allowed until after 2-month primary endpoint).

   - As recommended in ACC/AHA 2017 Guideline,2 subjects are to be taking one anti-hypertensive antagonizing the renin-angiotensin system, including ACE inhibitor, ARB or renin inhibitor. Second drug should either be a calcium channel blocker (amlodipine preferred) or a thiazide diuretic.
2. Stable antihypertensive medical regimen for at least 30 days.
3. Ambulatory mean daytime SBP ≥135 mmHg.
4. Ambulatory daytime SBP <170 and DBP <105 mmHg.
5. Office systolic SBP ≥140 mmHg and <180.

Exclusion Criteria:

1. History of non-compliance with medical care or medical treatments.
2. History of atrial fibrillation.
3. Pregnant (verified with a urine or blood pregnancy test), breast-feeding, or planning to become pregnant. Note that all premenopausal women will be screened for pregnancy (see section 4.7.4).
4. Office SBP ≥180 and DBP ≥110 mmHg.
5. Untreated urinary tract infection.
6. Renal collecting system is compromised, such that the subject cannot undergo routine cystoscopy and retrograde pyelogram, as exemplified by duplicated collecting system, i.e., two or more ipsilateral ureters.
7. Pre-existing hydronephrosis, presence of renal calculi or ectopic, pelvic or ptotic kidney(s).
8. Receiving dialysis treatment.
9. Renal transplant recipient.
10. Presence of only one kidney, or patients with dominant unilateral kidney function with one kidney split function less than 35%
11. Polycystic kidney disease.
12. Diabetes treated with SGLT2 inhibitor and/or GLP-1 agonist
13. Persistent albuminuria (urine with 30-300 mg albumin/g creatinine)
14. Focal sclerosing glomerulosclerosis.
15. On any of the following medications: clonidine, guanfacine, or methyldopa.
16. Known secondary causes of hypertension such as adrenal disease, renal artery stenosis, renovascular hypertension.
17. Evidence in medical history or at screening of hyperaldosteronism, defined as aldosterone/renin activity > 30 or aldosterone level >15 ng/dL
18. Glomerulonephritis or interstitial nephritis or eGFR <45 ml/min/1.73m2.
19. Type I diabetes mellitus.
20. Stenotic valvular heart disease for which reduction of blood pressure would be hazardous.
21. One or more episodes of orthostatic hypotension within the prior 6 months defined in section 6.6.2 as reduction of systolic blood pressure of ≥20 mmHg or diastolic blood pressure of ≥10 mm Hg within 3 minutes of standing.
22. Myocardial infarction, unstable angina, or stroke in the prior 6 months.
23. History of symptomatic heart failure
24. Echocardiographic evidence of dilated, infiltrative or hypertrophic cardiomyopathy or intracardiac mass.
25. Surgically correctable valvular heart disease.
26. Peripheral arterial disease manifest clinically by claudication or non-healing ulcers.
27. Any medical condition (including psychiatric disease) that would interfere with conducting the study or would not be in the best interest of the subject.
28. Prior diagnosis of pulmonary hypertension, use of chronic oxygen therapy or need for mechanical ventilation
29. Presence of severe obstructive sleep apnea not treated adequately by CPAP at screening.
30. On medications that affect blood pressure through off target effects, e.g., NSAIDs, steroids etc.
31. Uncorrected bleeding diathesis
32. Any clinical condition that can affect blood pressure or require the use of medications that can affect blood pressure (e.g., NSAIDs, steroids, cold remedies).
33. Life expectancy < 24 months for any reason (investigator determination).
34. Works night shifts.
35. Upper arm circumference > 20".
36. Subjects currently enrolled in another hypertension trial.
37. Subjects who previously received device therapy for hypertension, including renal denervation.
38. Subjects with a history of recurrent renal stones including episodes within the prior 6 months (subjects with first diagnosis of asymptomatic renal stone(s) at baseline/screening can be treated and rescreened at least one week following successful therapy of nephrolithiasis).
39. History of narcotic / opiate drug abuse
40. History of chronic pain syndrome receiving ongoing therapy with narcotic and/or opiate therapy
41. Active uroepithelial cancer
42. Artificial urinary sphincter or penile prosthesis implanted.
43. Planned medical procedures that could potentially interfere with measurement of blood pressure or assessment of any safety/effectiveness endpoints within 12 months of randomization
44. Conditions that could potentially interfere with accuracy of blood pressure measurements
45. Vulnerable subject populations (e.g., incarcerated or cognitively challenged adults).
46. Pre-existing urological abnormalities such as hydronephrosis, ureteral vesicular reflux (congenital or acquired), neoplasia, etc.
47. Urinary tract anomalies or primary (FSGS) or secondary (e.g., Diabetic nephropathy) renal disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2029-03-02 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness | 2 months post treatment
  effects of the device/procedure on 24-hour blood pressure control in addition to use of 2 antihypertensive medications

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Panoramic Health / Southwest Kidney Institute, PLC, Surprise, Arizona
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - DaVita Clinical Research, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No